CLINICAL TRIAL: NCT05125029
Title: Double Blind RCT to Evaluate the Effect of Botulinum Toxin in Raynaud Phenomenon
Brief Title: Botulinum Toxin in Raynaud's Phenomenon
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: American Society for Surgery of the Hand (Other)
Responsible Party: Principal Investigator, Paul A Ghareeb, MD, Assistant Professor of Surgery, Emory University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: STUDY00002359
Record Dates: First submitted 2021-10-26; First posted 2021-11-18 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-02

CONDITIONS: Raynaud Phenomenon
Keywords: Botulinum toxin; Raynaud Phenomenon refractory to treatment
MeSH Terms: conditions — Raynaud Disease | interventions — Botulinum Toxins

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Placebo (No Intervention): Prior to injection, patients will wait in a temperature controlled room for 30 minutes in order to allow time for normalization of baseline digital temperature. Once a patient is randomly selected via our randomization process, BT will be reconstituted by clinic nursing staff with sterile saline per manufacturer recommendations such that the investigating hand surgeon who will be performing the injection will be sufficiently blinded. After proper cleansing of the skin with alcohol swabs, BT will be sterilely administered percutaneously via a small-gauge needle and syringe into the base of each digit by the investigating hand surgeons within the Upper Extremity Division. The volar metacarpal head will be used as a standardized anatomic landmark for injection both to lessen the probability and magnitude of risk to deep structures of the hand as well as maximize probability of proper anatomic placement of the drug.
- 10 units of BT per digit (Active Comparator): Prior to injection, patients will wait in a temperature controlled room for 30 minutes in order to allow time for normalization of baseline digital temperature. Once a patient is randomly selected via our randomization process, BT will be reconstituted by clinic nursing staff with sterile saline per manufacturer recommendations such that the investigating hand surgeon who will be performing the injection will be sufficiently blinded. After proper cleansing of the skin with alcohol swabs, BT will be sterilely administered percutaneously via a small-gauge needle and syringe into the base of each digit by the investigating hand surgeons within the Upper Extremity Division. The volar metacarpal head will be used as a standardized anatomic landmark for injection both to lessen the probability and magnitude of risk to deep structures of the hand as well as maximize probability of proper anatomic placement of the drug.
  Interventions: Drug: Botulinum toxin
- 20 units of BT per digit (Active Comparator): Prior to injection, patients will wait in a temperature controlled room for 30 minutes in order to allow time for normalization of baseline digital temperature. Once a patient is randomly selected via our randomization process, BT will be reconstituted by clinic nursing staff with sterile saline per manufacturer recommendations such that the investigating hand surgeon who will be performing the injection will be sufficiently blinded. After proper cleansing of the skin with alcohol swabs, BT will be sterilely administered percutaneously via a small-gauge needle and syringe into the base of each digit by the investigating hand surgeons within the Upper Extremity Division. The volar metacarpal head will be used as a standardized anatomic landmark for injection both to lessen the probability and magnitude of risk to deep structures of the hand as well as maximize probability of proper anatomic placement of the drug.
  Interventions: Drug: Botulinum toxin

INTERVENTIONS:
Drug: Botulinum toxin — Botulinum toxin is a neurotoxic protein produced by the bacterium Clostridium botulinum that prevents the release of the neurotransmitter acetylcholine from the neuromuscular junction, thereby preventing muscular contraction. Eligible subjects will be randomized 1:1:1 into three different groups: 1) placebo 2) 10 Units of BT injected per digit and 3) 20 units of BT injected per digit.
  Arms: 10 units of BT per digit; 20 units of BT per digit

SUMMARY:
Raynaud's Phenomenon (RP) is the most common vasospastic disorder encountered by hand surgeons with an estimated prevalence of 5% in the general population. It's manifestations are broad, and can range from minor to severe. Sometimes it can be refractory to treatments. The goal of this study is to evaluate the efficacy of Botulinum toxin (BT) in the treatment of treatment refractory RP by objective and subjective measures.

DETAILED DESCRIPTION:
Raynaud's Phenomenon (RP) is the most common vasospastic (i.e. conditions where small blood vessels near the surface of the skin have spasms that limit blood flow) disorder encountered by hand surgeons with an estimated prevalence of 5% in the general population. The clinical manifestations are broad, and can range from minor pain, cold sensitivity and color changes to impaired hand function, intolerable pain and tissue loss/digital ulceration. Treatment algorithms include activity modification and medical therapies. However, refractory RP can warrant surgical intervention, such as peri-arterial sympathectomy, of which has significant associated morbidity. While the exact mechanism is still being elucidated, several retrospective reviews have demonstrated efficacy of BT in the treatment of RP. Specifically, increases in post treatment perfusion have been demonstrated and clinical evidence of improvement in pain scores and tissue loss are reported. However, the literature varies in regard to injection technique (location and dose) and duration of action.

The goal of this study is to evaluate the efficacy of BT in the treatment of treatment refractory RP by objective and subjective measures. This study will perform a single-site double-blinded, randomized, placebo-controlled trial evaluating two different doses of BT (10 units and 20 units) injected into each patient's fingers of both hands versus injection of a normal saline control, given that there is currently no widely accepted standard of care for the treatment of BT. Following injection, patients will be evaluated in regular intervals to assess for impact on finger temperature, oxygenation, patient reported outcome measures (PROMs), and effect on tissue loss.

The study will take place under Emory University School of Medicine, specifically the Upper Extremity Division. Patients may also be originally seen under the Rheumatology Division and subsequently referred to the Upper Extremity Division for study participation. In total, the study aims to recruit 36 patients. There will be no outside recruitment or advertisement materials. With this research study, the study team seeks to establish a standardized injection technique and dosage for this disease and to determine duration of symptom alleviation.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older
* Patients with moderate to severe RP that is not controlled after 3 months of standard medical therapy as prescribed by a Rheumatologist, or severe RP with evidence of tissue loss.

Exclusion Criteria:

* Patients under the age of 18
* Patients who have previously undergone treatment with BT for RP within the past year
* Patients with active infection at the treatment site (active infection defined as cellulitis, purulence, fever, chills, or presence of elevated inflammatory markers, ie. WBC, ESR, CRP)
* Patients who have undergone prior digital sympathectomy surgery for RP
* Patients who have recently altered their medical regimen for RP within the past 4 weeks
* Patients with allergy or contraindication to BT injection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2022-02-10 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Change in finger temperature measure | Baseline, 4 weeks, 12 weeks, 24 weeks post injection
  Temperature of the each finger on each hand will be evaluated pre-treatment and at regular follow up intervals baseline, 4 weeks, 12 weeks, 24 weeks post injection
Change in tissue Oximetry measure for each finger | Baseline, 4 weeks, 12 weeks, 24 weeks post injection
  Tissue Oximetry of each finger on each hand will be recorded on each digit prior to treatment and at the allotted follow up intervals.

SECONDARY OUTCOMES:
Changes in Raynaud Condition Score | Performed at 4 weeks, 12 weeks, 16 weeks, 20 weeks, and 24 weeks. Week 16 and week 20 measurements will be performed via telephone interview.
  The Raynaud's Condition Score (RCS) is a validated outcome measure used to assess the level of difficulty experienced due to RP each day (anchored from "no difficulty" to "extreme difficulty").
Changes in Visual Analog Scale (VAS) pain score | Performed at 4 weeks, 12 weeks, 16 weeks, 20 weeks, and 24 weeks. Week 16 and week 20 measurements will be performed via telephone interview.
  The visual analogue scale or visual analog scale (VAS) is a psychometric response scale which can be used in questionnaires. It is a measurement instrument for subjective characteristics or attitudes that cannot be directly measured. When responding to a VAS item, respondents specify their level of agreement to a statement by indicating a position along a continuous line between two end-points.
Changes in PROMIS Pain Interference scale | Performed at 4 weeks, 12 weeks, 16 weeks, 20 weeks, and 24 weeks. Week 16 and week 20 measurements will be performed via telephone interview.
  PROMIS Pain Interference (PROMIS-PI) scale measures the extent to which pain hinders an individual's engagement with physical, mental, cognitive, emotional, recreational, and social activities.
Changes in Hand subjectivity value | Performed at 4 weeks, 12 weeks, 16 weeks, 20 weeks, and 24 weeks. Week 16 and week 20 measurements will be performed via telephone interview.
  Patients will provide ratings of their subjective hand function from 0 to 100
Changes in QUICK Dash assessment | Performed at 4 weeks, 12 weeks, 16 weeks, 20 weeks, and 24 weeks. Week 16 and week 20 measurements will be performed via telephone interview.
  The Quick DASH uses 11 items to measure physical function and symptoms in people with any or multiple musculoskeletal disorders of the upper limb. It is scored in two components: the disability/symptom section (11 items, scored 1-5) and the optional high performance sport/music or work modules (four items, scored 1-5).

CONTACTS AND LOCATIONS:
Overall Officials: Paul A Ghareeb, MD, Principal Investigator — Emory University
Locations (1):
- Emory University Hospital, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: No
No individual de-identified participant data will be shared